CLINICAL TRIAL: NCT05448495
Title: Posterior Transversus Abdominis Plane Block Versus Erector Spinae Plane Block as a Part of Multimodal Analgesia in Patients Undergoing Percutaneous Nephrolithotomy. A Prospective Randomized Clinical Trial
Brief Title: Posterior Transversus Abdominis Plane Block Versus Erector Spinae Plane Block as a Part of Multimodal Analgesia in Patients Undergoing Percutaneous Nephrolithotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, FATMA NABIL AHMED MOHAMED, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Posterior TAPB versus ERSPB
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Analgesia
Keywords: Percutaneous nephrolithotomy; Erector spinae plane block; Transversus abdominis plane block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior TAP block (Experimental)
  Interventions: Other: Posterior TAP block
- ESPB (Active Comparator)
  Interventions: Other: ESPB

INTERVENTIONS:
Other: Posterior TAP block — Using high-frequency linear ultrasound probe, a total volume of 24 ml (20 ml isobaric bupivacaine 0.5% + 2 ml dexmedetomidine [0.5 mcg\kg] + 2ml dexamethasone [0.1mg\kg)] will be injected at the plane between internal oblique and transversus abdominis near the aponeurosis at the posterior axillary line.
  Other Names: Posterior transversus abdominis plane block
  Arms: Posterior TAP block
Other: ESPB — Using high-frequency linear ultrasound probe, a total volume of 24 ml (20 ml isobaric bupivacaine 0.5% + 2 ml dexmedetomidine [0.5 mcg\kg] + 2ml dexamethasone [0.1mg\kg)] will be injected at T9 erector spinae plane
  Other Names: Erector spinae plane block
  Arms: ESPB

SUMMARY:
To compare the analgesic efficacy of posterior TAP block versus ESPB after PCNL surgery. The hypothesis is that posterior TAP block, as a part of multimodal analgesia, will reduce pain and opioid consumption like ESPB

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is currently the gold standard for treatment of patients with large and complex renal calculi because it is less invasive than open surgery. The sources of acute pain after PCNL are visceral pain originating from kidneys and ureters, and somatic pain from the site incision. PCNL is usually done in 10th to 11th intercostal space or in the subcostal area. Complete blockade of unilateral spinal nerves from T10 to L2 can provide sufficient analgesia during PCNL. This can be achieved by several regional techniques such as thoracic paravertebral block, transversus abdominis plane (TAP) block, erector spinae plane block (ESPB).

ESPB is an interfascial block which can provide wide sensory blockade from T2-4 to L1-2 that was first described in 2016. ESPB can be performed by injecting the local anesthetic in the deep interfascial plane of the erector spinae muscle with nearly one dermatome for each 3.4 ml of the injected volume. This allows ESPB to provide both visceral and somatic analgesia. TAP block is a regional injection of a local anesthetic agent between the transversus abdominis and internal oblique muscle planes. TAP block affects the sensory nerves of the anterolateral abdominal wall (T6-L1). Various technical modifications in TAP block have been described including lateral, posterior, subcostal, and continuous catheter techniques. The posterior approach should be the preferred technique in clinical practice as it provides longer somatic and visceral analgesia that are not offered with the lateral approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for PCNL under general anesthesia
* ASA status I-II

Exclusion Criteria:

1. Contraindications to regional block (coagulopathy, infection at the needle insertion site or known allergy to amide local anesthetics)
2. Patient who has difficulty understanding the study protocol or patient refusal.
3. Chronic respiratory disease patients.
4. Diabetic patients.
5. Body mass index (BMI) > 30 Kg/m2
6. Routine corticosteroids, pain medication, or anticonvulsant.
7. Psychiatric diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
The time to first call rescue analgesia | From end of surgery till 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided